CLINICAL TRIAL: NCT01920945
Title: OnabotulinumtoxinA for the Treatment of New Daily Persistent Headache: an Open Label Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult enrollment
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLERGAN-13-002
Record Dates: First submitted 2013-08-07; First posted 2013-08-12 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: New Daily Persistent Headache
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OnabotulinumtoxinA (Experimental)
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: OnabotulinumtoxinA — 155 units of OnabotulinumtoxinA, will be injected into 31 sites in the head and neck every 12 weeks for a total of 24 weeks using a sterile 30-gauge, 0.5 inch needle as 0.1 mL (5 Units) injections per each site. Injections will be divided across seven specific head/neck muscle areas (corrugator, procerus, frontalis, temporalis, suboccipital, splenius capitus and medial/lateral occipital, and trapezius).
  Other Names: Botox

SUMMARY:
The purpose of this study is to evaluate the effect of BOTOX® (OnabotulinumtoxinA) on the number of headache days in patients with New Daily Persistent Headache (NDPH). NDPH is a benign form of chronic daily headache that comes in two forms: one that resolves on its own after months to years, or one that is difficult to treat and does not respond to preventive or abortive medications. Some patients experience migrainous features such as nausea, vomiting, photophobia, or phonophobia. BOTOX®, a treatment approved for chronic migraine, will be injected into specific muscles of the head and neck area by your study doctor, to evaluate its effectiveness in reducing or relieving NDPH days or severity. BOTOX has not been approved for NDPH and this is the first time it will be used for treatment of NDPH. All participants in this study will only receive BOTOX® and no other study drug.

ELIGIBILITY:
Inclusion Criteria:

Subjects aged 18 or older, male or female of any race with the diagnosis of NDPH meeting International Classification of Headache Disorders (ICHD-2) criteria will be included in the study. The criteria is as follows:

A. Persistent headache fulfilling criteria B and C B. Distinct and clearly remembered onset, with pain becoming continuous and unremitting within 24 hours C. Present for >3 months D. Not better accounted for by another ICHD-3 diagnosis

Exclusion Criteria:

1. Those with relevant physical or psychological illness, particularly conditions that might put them at risk if exposed to OnabotulinumtoxinA (myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other neuromuscular disease).
2. Diagnosis of other primary/secondary headache disorder.
3. Psychiatric disorders that could interfere with study participation.
4. Subjects who abuse drugs, including headache treatments and alcohol (DSM IV criteria).
5. Those allergic to compounds similar to the study medication.
6. Those who are pregnant or breastfeeding, or who do not use adequate contraceptive methods.
7. Those who have had any prior exposure to any botulinum toxin serotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
change from baseline in frequency of headache days | 29 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Roosevelt Hospital Headache Institute, New York, New York, United States